CLINICAL TRIAL: NCT04909814
Title: Colposcopic Impression in a Birth Cohort Previously Eligible for HPV-vaccination
Status: Completed | Type: Observational
Sponsor: Falu Hospital (Other)
Responsible Party: Principal Investigator, Hanna Sahlgren, Principal Investigator, Falu Hospital
Other Study IDs: 2018/535-31/1
Record Dates: First submitted 2021-05-27; First posted 2021-06-02 (Actual); Last update posted 2021-06-07 (Actual); Status verified 2021-06

CONDITIONS: HPV; Cervical Cancer
Keywords: colposcopy
MeSH Terms: conditions — Uterine Cervical Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Vaccinated women with positive screening test: All women in one Swedish county taking their first screening test within the organized cervical screening program
  Interventions: Biological: The performance of colposcopy in vaccinated women

INTERVENTIONS:
Biological: The performance of colposcopy in vaccinated women — Evaluating the performance of colpscopy in HPV vaccinated women by comparing vaccinated and unvaccinated women taking their first test within the organized screening program

SUMMARY:
Women were invited to attend colposcopy within two-four months after a positive screening test (two consecutive screening tests indicating low-grade squamous intraepithelial lesions (LSIL) and HPV positivity or a single screening test indicating high grade squamous intraepithelial lesions (HSIL)), according to national guidelines

DETAILED DESCRIPTION:
To describe the source population, the overall number of invitations and tests taken in the region during the study period were retrieved from the Swedish National Cervical Screening Registry (NKCx), which has an almost 100% coverage of screening history in Sweden since 1993.

Women were invited to attend colposcopy within two-four months after a positive screening test (two consecutive screening tests indicating low-grade squamous intraepithelial lesions (LSIL) and HPV positivity or a single screening test indicating high grade squamous intraepithelial lesions (HSIL)), according to national guidelines. All colposcopies were performed in 2018 and 2019 at the Department of Obstetrics and Gynecology, Falun Hospital, by a specialist in Obstetrics and Gynecology. Digital imaging ensured the possibility of subsequent re-review by an expert colposcopist at the Karolinska University Hospital. The colposcopies consisted of a microscopic evaluation of the uterine cervix including punch biopsies as well as endocervical sampling with liquid based cytology (LBC). In the absence of visible colposcopic lesions, random biopsies at 6 and 12 o´clock were taken to ensure histopathological confirmation in all women. Women with colposcopic and/or histopathologic findings that required treatment underwent excision (conization) according to national guidelines. The consultation also included questions on medical history according to a protocol designed for the study.

Analysis of histopathology and cytology was performed at the Department of Pathology, Falun Hospital. An LBC sample was analyzed for the presence of 14 high risk HPV (hrHPV) genotypes and cytology. HPV samples were tested at the Department of Laboratory Medicine, Falun Hospital, using amplification of target DNA by the Polymerase Chain Reaction (PCR) and nucleic acid hybridization (Cobas 4800, Roche Molecular Systems). LBC samples positive for high risk types other than HPV 16/18, were sent for further genotyping to the Center for Cervical Cancer Prevention at the Karolinska University Laboratory Huddinge.

Information on vaccination status was retrieved through linkage to the National HPV Vaccination Register (SVEVAC), an informed consent-based register in operation since the introduction of HPV vaccination In Sweden, and data was further complemented by linkage to the Prescribed Drug Register (PDR), a mandatory register on dispensed prescriptions in Sweden in operation since July 2005. All women were asked about their vaccination status after the colposcopic examination had been performed, and linkage to SVEVAC and PDR was run after all study colposcopies and laboratory analysis had been completed. Hence, vaccination status was blinded to the colposcopists, pathologists, and laboratory staff.

ELIGIBILITY:
Inclusion Criteria:

- HPV-vaccinated women Women taking their first test within the organized cervical screening program at age 23 Women residing in one Swedish county

Exclusion Criteria:

Women who were hysterectomized, Women who died Women who moved

-

Ages: 22 Years to 26 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Only women go through colpsocopy
Study Population: Women were invited to attend colposcopy within two-four months after a positive screening test (two consecutive screening tests indicating low-grade squamous intraepithelial lesions (LSIL) and HPV positivity or a single screening test indicating high grade squamous intraepithelial lesions (HSIL)), according to national guidelines
Sampling Method: Probability Sample
Enrollment: 160 (Actual)
Dates: Start 2018-03-14 (Actual); Primary Completion 2019-10-15 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Performance of the Swedscore colposcopy scale in HPV-vaccinated women | 1 year
  Positive predictive value of colposcopy for high grade lesions in HPV-vaccinated women

CONTACTS AND LOCATIONS:
Overall Officials: Hanna I Sahlgren, md, Principal Investigator — RCC; Miriam K Elfström, phd, Principal Investigator — RCC
Locations (1):
- Falu Lasarett, Falun, Dalarna County, Sweden

IPD SHARING:
Plan to Share IPD: Yes
On demand
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: 3 years
Access Criteria: Contact Principal investigator

REFERENCES:
- [Derived] Sahlgren HAI, Elfgren K, Sparen P, Elfstrom MK. Colposcopic performance in a birth cohort previously eligible for human papillomavirus vaccination. Am J Obstet Gynecol. 2022 May;226(5):704.e1-704.e9. doi: 10.1016/j.ajog.2021.11.1372. Epub 2021 Dec 23. PMID 34954217